CLINICAL TRIAL: NCT03538301
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, Biological Activity, and PK of ND-L02-s0201 in Subjects With Idiopathic Pulmonary Fibrosis (IPF)
Brief Title: JUNIPER: A Phase 2 Study to Evaluate the Safety, Biological Activity, and PK of ND-L02-s0201 in Subjects With IPF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nitto Denko Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ND-L02-s0201-005
Record Dates: First submitted 2018-05-02; First posted 2018-05-29 (Actual); Results first posted 2023-12-11 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-11

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose Level 1 (Experimental): ND-L02-s0201 45mg
  Interventions: Drug: ND-L02-s0201 (Low Dose)
- Dose Level 2 (Experimental): ND-L02-s0201 90mg
  Interventions: Drug: ND-L02-s0201 (High Dose)
- Placebo (Placebo Comparator): Control Arm
  Interventions: Other: Other: Placebo

INTERVENTIONS:
Drug: ND-L02-s0201 (Low Dose) — Intravenous administration every 2 weeks
  Other Names: 45mg
  Arms: Dose Level 1
Drug: ND-L02-s0201 (High Dose) — Intravenous administration every 2 weeks
  Other Names: 90mg
  Arms: Dose Level 2
Other: Other: Placebo — Saline
  Arms: Placebo

SUMMARY:
A phase 2, randomized, double-blind, placebo-controlled, multicenter study to evaluate the safety, tolerability, biological activity, and pharmacokinetics (PK) of ND-L02-s0201 for Injection in subjects with IPF.

DETAILED DESCRIPTION:
All subjects were treated with ND-L02-s0201 or placebo for 24 weeks (a total of 12 doses). Subject's participation in the study was approximately 40 weeks including a Screening and Baseline period of up to 6 weeks, a treatment period of 24 weeks (including the 2 weeks after the last study treatment), and a follow-up period of 10 weeks after End-of-Treatment (EOT).

ELIGIBILITY:
Inclusion Criteria:

* Forced vital capacity (FVC) ≥ 45% of predicted.
* Diffusion capacity of the lung for carbon monoxide (DLco) corrected for hemoglobin ≥ 30% of predicted value
* Ratio of forced expiratory volume in 1 second (FEV1) to FVC ≥ 0.70.

Exclusion Criteria:

* Best, acceptable FVC from separate screening spirometry that differ by ≥ 200 mL.
* Respiratory exacerbation(s) or hospitalization for IPF exacerbation within 3 months before screening.
* Anticipated to receive a lung transplant during the subject's participation in the study.
* Active smoker or smoking cessation within 12 weeks before screening.
* Malignancy within the last 5 years, with the exception of curable cancer that has received adequate treatment.
* Evidence of any unstable or untreated, clinically significant disease or condition that, in the opinion of the Investigator, might confound the interpretation of the study or place the subject at increased risk.
* Treatment with high dose corticosteroids, cytotoxic agents, unapproved IPF targeted therapy, and cytokine modulating agents within 8 weeks or 5 half-lives (whichever is longer) before screening
* Participation in an investigational study with the last dose of investigational product occurring within 8 weeks or 5 half-lives (whichever is longer) before screening.
* Pregnant or breastfeeding.
* Medical history of infection with HIV, hepatitis B, or hepatitis C.
* History of alcohol abuse and/or dependence within the last 2 years.
* History within the last 2 years of significant mental illness, or physical dependence on any opioid or illicit drugs.

Other protocol defined inclusion/exclusion criteria could apply.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2022-08-24 (Actual); Study Completion 2022-08-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nitto Denko Corporation, Study Director — Nitto Denko Corporation
Locations (33):
- United States (21):
  - Banner-University Medical Center Tucson Campus, Tucson, Arizona
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Amicis Research Center, Northridge, California
  - University of California, San Francisco, Medical Center at Parnassus, San Francisco, California
  - Mayo Clinic Florida, Jacksonville, Florida
  - Central Florida Pulmonary Group, PA, Orlando, Florida
  - Emory University, Atlanta, Georgia
  - Loyola University Medical Center, Maywood, Illinois
  - OSF HealthCare Saint Francis Medical Center, Peoria, Illinois
  - Norton Clinical Research Group, Louisville, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Minnesota Medical School, Minneapolis, Minnesota
  - Dartmouth-Hitchcock Medical Center (DHMC), Lebanon, New Hampshire
  - Duke University Hospital, Durham, North Carolina
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - UT Southwestern Medical Center, Dallas, Texas
  - UT Health San Antonio: First Outpatient Research Unit, San Antonio, Texas
  - University of Utah Health, Salt Lake City, Utah
  - University of Washington, Seattle, Washington
- Germany (6):
  - Universitatsklinikum Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Thoraxklinik-Heidelberg gGmbH, Heidelberg, Baden-Wurttemberg
  - Justus-Liebig-Universitaet Giessen, Giessen, Hesse
  - Lungenfachklinik Immenhausen, Immenhausen, Hesse
  - Medizinische Hochschule Hannover (MHH), Hanover, Lower Saxony
  - Ruhrlandklinik, Universitatmedzin Essen, Essen, North Rhine-Westphalia
- Japan (5):
  - National Hospital Organization Himeji Medical Center, Himeji-Shi, Hyōgo
  - National Hospital Organization Ibarakihigashi National Hospital, Naka-gun, Ibaraki
  - Kanagawa Cardiovascular and Respiratory Center, Yokohama, Kanagawa
  - National Hospital Organization Kinki-chuo Chest Medical Center, Osaka, Sakai-shi
  - Tosei General Hospital, Aichi, Seto-shi
- Royal Papworth Hospital NHS Foundation Trust, Cambridge, Cambridgeshire, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Diagnosis of idiopathic pulmonary fibrosis within 5 years before Visit 1a, confirmed by the Principal Investigator (PI) using American Thoracic Society (ATS)/European Respiratory Society (ERS)/Japanese Respiratory Society (JRS)/Latin American Thoracic Association (ALAT) guidelines
Groups:
- Placebo: Intravenous placebo infusion every 2 weeks (± 4 days for Visit 3 or ± 7 days for Visits 4 to 13, ensuring a minimum of 7 days between each dose) for a total of 12 doses.
- ND-L02-s0201 45 mg: ND-L02-s0201: 45 mg intravenous administration every 2 weeks (± 4 days for Visit 3 or ± 7 days for Visits 4 to 13, ensuring a minimum of 7 days between each dose) for a total of 12 doses.
- ND-L02-s0201 90 mg: ND-L02-s0201: 90 mg intravenous administration every 2 weeks (± 4 days for Visit 3 or ± 7 days for Visits 4 to 13, ensuring a minimum of 7 days between each dose) for a total of 12 doses.
Period: Overall Study
Arm/Group | Placebo | ND-L02-s0201 45 mg | ND-L02-s0201 90 mg
Started | 42 | 41 | 40
Completed | 31 | 29 | 28
Not Completed | 11 | 12 | 12
Not completed — Adverse Event | 1 | 4 | 4
Not completed — Death | 1 | 1 | 0
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Terminated Early from the Study due to COVID-19 Impact | 9 | 6 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | ND-L02-s0201 45 mg | ND-L02-s0201 90 mg | Total
Number analyzed (Participants) | 42 | 41 | 40 | 123
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at screening
  years | 68.7 (6.16) | 68.9 (6.22) | 69.2 (6.53) | 68.9 (6.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 6 | 18
  Male | 37 | 34 | 34 | 105
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 2 | 4 | 11
  Not Hispanic or Latino | 37 | 39 | 36 | 112
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 7 | 10 | 7 | 24
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 1 | 3
  White | 34 | 29 | 31 | 94
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1 | 2
Smoking History [Count of Participants; unit: Participants]
  Yes | 26 | 27 | 26 | 79
  No | 16 | 14 | 14 | 44
Background Standard of Care [Count of Participants; unit: Participants]
  Nintedanib | 17 | 17 | 16 | 50
  Pirfenidone | 15 | 14 | 14 | 43
  None | 10 | 10 | 10 | 30
Height [Mean (Standard Deviation); unit: centimeters] | 172.399 (6.5281) | 172.316 (10.5278) | 171.519 (9.2947) | 172.085 (8.8564)
Weight [Mean (Standard Deviation); unit: kilograms] | 85.579 (15.4326) | 84.234 (19.0174) | 82.255 (17.6139) | 84.050 (17.3109)
Body mass index (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 28.765 (4.7625) | 28.093 (4.3072) | 27.780 (4.5129) | 28.221 (4.5151)
Body mass index group [Count of Participants; unit: Participants] — Category ranges are in kg/m^2.
  Participants
    Underweight (below 18.5) | 0 | 0 | 0 | 0
    Normal (18.5 - 24.9) | 12 | 11 | 10 | 33
    Overweight (25 - 29.9) | 15 | 17 | 22 | 54
    Obese (30 and above) | 15 | 13 | 8 | 36
Baseline Pulse Oximetry (%) [Mean (Standard Deviation); unit: % of oxygen saturated hemoglobin] | 96.5 (2.11) | 96.6 (1.99) | 96.9 (1.93) | 96.7 (2.00)
Baseline Forced Vital Capacity [Mean (Standard Deviation); unit: litres] | 2.861 (0.7214) | 3.012 (0.6866) | 2.890 (0.7562) | 2.921 (0.7188)
Baseline Percent Predicted Forced Vital Capacity (%) [Mean (Standard Deviation); unit: % of total normal FVC] | 73.943 (17.0078) | 79.319 (14.9940) | 76.658 (18.1270) | 76.618 (16.7595)
Baseline Forced Expiratory Volume in 1 second [Mean (Standard Deviation); unit: litres] | 2.270 (0.5603) | 2.380 (0.5345) | 2.274 (0.5890) | 2.308 (0.5592)
Baseline Percent Predicted Forced Expiratory Volume [Mean (Standard Deviation); unit: % of normal FEV] | 76.890 (17.8868) | 81.959 (14.8182) | 78.766 (17.6653) | 79.190 (16.8442)
Baseline Ratio of Forced Expiratory Volume in 1 second/Forced Vital Capacity [Mean (Standard Deviation); unit: ratio] | 0.795 (0.0501) | 0.794 (0.0383) | 0.787 (0.0450) | 0.792 (0.0445)
Baseline Diffusion Capacity of the Lung for Carbon Monoxide Corrected for Hemoglobin [Mean (Standard Deviation); unit: mL/min/mmHg] | 12.574 (3.9023) | 12.972 (3.6453) | 12.391 (3.3503) | 12.647 (3.6223)
Baseline Hemoglobin Corrected percent predicted DLCO [Mean (Standard Deviation); unit: % of normal DLCO] — DLCO = diffusion capacity of the lung for carbon monoxide
  % of normal DLCO | 51.762 (14.7970) | 53.739 (13.1901) | 51.914 (12.6957) | 52.471 (13.5264)
Eligibility Criteria Based on high resolution computed tomography [Count of Participants; unit: Participants] — Participants were staged based on the presence or absence of a usual interstitial pneumonia (UIP) pattern on chest HRCT scans assessments.
  The diagnosis of IPF will be confirmed by the PI using ATS/ERS/JRS/ALAT consensus criteria (Raghu et al, 2011: https://www.atsjournals.org/doi/full/10.1164/rccm.2009-040GL).
  Please refer to protocol section 11.2.5
  Participants
    Definite UIP | 30 | 26 | 22 | 78
    Consistent with UIP | 6 | 10 | 11 | 27
    Possible UIP | 1 | 0 | 0 | 1
    Inconsistent with UIP | 5 | 5 | 7 | 17
    Unknown | 0 | 0 | 0 | 0
Duration of idiopathic pulmonary fibrosis [Mean (Standard Deviation); unit: months] | 28.227 (17.4342) | 24.678 (16.3543) | 27.272 (15.7152) | 26.734 (16.4642)
GAP IPF Stage [Count of Participants; unit: Participants] — The GAP IPF stage for each subject was calculated by adding up the points assigned to categories I, II, and III, where stage I is the better and stage III is the worst.
  gender (G); age (A); baseline FVC,% predicted; and baseline DLco, % predicted
  Refer to SAP- Appendix 1: GAP Algorithm for IPF Stage and Predicted Mortality
  Participants
    I (0 to 3 points. This stage has the lowest risk of mortality | 24 | 29 | 25 | 78
    II (4 to 5 points. This stage has a moderate risk of mortality) | 17 | 11 | 15 | 43
    III (6 to 8 points. This stage has the highest risk of mortality) | 1 | 1 | 0 | 2
Risk of Mortality at 1-year [Mean (Standard Deviation); unit: risk ratio] — The risk of mortality (1-, 2-, and 3-year risk) will be derived based on baseline data at the start of the treatment period using the Gender, Age, and Physiology (GAP) methodology. Risk of mortality will be derived using the algorithm listed in SAP- Appendix 1: GAP Algorithm for IPF Stage and Predicted Mortality.
  risk ratio | 14.726 (7.1570) | 12.584 (4.9287) | 13.930 (6.0984) | 13.753 (6.1532)
Risk of Mortality at 2-year [Mean (Standard Deviation); unit: risk ratio] — The risk of mortality (1-, 2-, and 3-year risk) will be derived based on baseline data at the start of the treatment period using the Gender, Age, and Physiology (GAP) methodology. Risk of mortality will be derived using the algorithm listed in SAP- Appendix 1: GAP Algorithm for IPF Stage and Predicted Mortality.
  risk ratio | 28.505 (12.5204) | 24.922 (9.0103) | 27.233 (11.0164) | 26.897 (10.9697)
Risk of Mortality at 3-year [Mean (Standard Deviation); unit: risk ratio] — The risk of mortality (1-, 2-, and 3-year risk) will be derived based on baseline data at the start of the treatment period using the Gender, Age, and Physiology (GAP) methodology. Risk of mortality will be derived using the algorithm listed in SAP- Appendix 1: GAP Algorithm for IPF Stage and Predicted Mortality.
  risk ratio | 40.335 (15.9727) | 36.014 (11.9575) | 38.869 (14.4372) | 38.418 (14.2311)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Discontinuing Study Treatment Due to TEAEs
Description: The number of participants with TEAEs leading to discontinuation from the study treatment. The Safety Population (including all participants who received at least one dose of study treatment) is presented.
  TEAE = treatment-emergent adverse event
Time Frame: Change in the incidence and severity of adverse events related to study treatment from baseline to 24 weeks
Population: Safety Population (includes all participants who received at least one dose of study treatment)
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | ND-L02-s0201 45 mg | ND-L02-s0201 90 mg
Number analyzed (Participants) | 42 | 41 | 40
Participants | 1 | 3 | 4

2. Secondary Outcome: Rate of Decline in FVC From Baseline to Week 24
Description: Slope in FVC from Baseline to Week 24 (measured in L/week). The intent-to-treat population (any randomized participants with treatment assignment according to the planned randomization) is presented.
  Slope and standard error are presented. The slope is approximated as least square mean/24 weeks.
  FVC = forced vital capacity
Time Frame: Baseline to Week 24
Population: ITT Population (include any randomized participants with treatment assignment according to the planned randomization)
Measure: Mean (Standard Error); unit: litres/week
Arm/Group | Placebo | ND-L02-s0201 45 mg | ND-L02-s0201 90 mg
Number analyzed (Participants) | 42 | 41 | 40
litres/week | -0.003366 (0.0014272) | -0.007519 (0.0015285) | -0.005478 (0.0015400)
Statistical Analysis 1: Comparison: Placebo vs ND-L02-s0201 45 mg; Slope in FVC (L/week) in the 45 mg cohort versus placebo; Test type: Superiority; p = 0.049, random coefficient model; Slope = -0.004153, 95% CI 2-sided [-0.008284 to -0.000021]
Statistical Analysis 2: Comparison: Placebo vs ND-L02-s0201 90 mg; Slope in FVC (L/week) in the 90 mg cohort versus placebo; Test type: Superiority; p = 0.316, random coefficient model; Slope = -0.002112, 95% CI 2-sided [-0.006260 to 0.002036]

3. Secondary Outcome: Rate of Decline in ppFVC From Baseline to Week 24
Description: Slope in ppFVC from Baseline to Week 24 (measured in %/week). The intent-to-treat population (any randomized participants with treatment assignment according to the planned randomization) is presented.
  Slope and standard error are presented. The slope is approximated as least square mean/24 weeks.
  ppFVC = percent predicted forced vital capacity
Time Frame: Baseline to Week 24
Population: ITT Population (include any randomized participants with treatment assignment according to the planned randomization)
Measure: Mean (Standard Error); unit: %/week
Arm/Group | Placebo | ND-L02-s0201 45 mg | ND-L02-s0201 90 mg
Number analyzed (Participants) | 42 | 41 | 40
%/week | -0.096455 (0.0373658) | -0.187694 (0.0400588) | -0.136051 (0.0403636)
Statistical Analysis 1: Comparison: Placebo vs ND-L02-s0201 45 mg; Test type: Superiority; p = 0.098, random coefficient model; Slope = -0.091238, 95% CI 2-sided [-0.199456 to 0.016979]
Statistical Analysis 2: Comparison: Placebo vs ND-L02-s0201 90 mg; Test type: Superiority; p = 0.473, random coefficient model; Slope = -0.039596, 95% CI 2-sided [-0.148248 to 0.069056]

4. Secondary Outcome: Absolute and Relative Change in FVC (L) From Baseline to Week 24
Description: Absolute and Relative Change in FVC (L) from Baseline to Week 24. The intent-to-treat population (any randomized participants with treatment assignment according to the planned randomization) is presented.
  FVC = forced vital capacity
Time Frame: Baseline to Week 24
Measure: Least Squares Mean (Standard Error); unit: litres
Arm/Group | Placebo | ND-L02-s0201 45 mg | ND-L02-s0201 90 mg
Number analyzed (Participants) | 42 | 41 | 40
litres
  Baseline FVC (L) | 2.8754 (0.11079) | 3.0242 (0.11207) | 2.9032 (0.11328)
  Week 24 FVC (L) | 2.7946 (0.10946) | 2.8438 (0.11144) | 2.7717 (0.11253)
  Change from Baseline to Week 24 in FVC (L) | -0.0808 (0.03425) | -0.1805 (0.03668) | -0.1315 (0.03696)
Statistical Analysis 1: Comparison: Placebo vs ND-L02-s0201 45 mg; Change from Baseline to Week 24 in FVC (L) in the 45 mg cohort versus placebo; Test type: Superiority; p = 0.049, random coefficient model; Mean Difference (Final Values) = -0.0997, 95% CI 2-sided [-0.1988 to -0.0005]
Statistical Analysis 2: Comparison: Placebo vs ND-L02-s0201 90 mg; Change from Baseline to Week 24 in FVC (L) in the 90 mg cohort versus placebo; Test type: Superiority; p = 0.316, random coefficient model; Mean Difference (Final Values) = -0.0507, 95% CI 2-sided [-0.1502 to 0.0489]

5. Secondary Outcome: Percent Change in FVC From Baseline to Week 24
Description: Percent Change in FVC from Baseline to Week 24. The intent-to-treat population (any randomized participants with treatment assignment according to the planned randomization) is presented.
  FVC = forced vital capacity
Time Frame: Baseline to Week 24
Population: ITT Population (include any randomized participants with treatment assignment according to the planned randomization)
Measure: Least Squares Mean (Standard Error); unit: percentage
Arm/Group | Placebo | ND-L02-s0201 45 mg | ND-L02-s0201 90 mg
Number analyzed (Participants) | 42 | 41 | 40
percentage | -3.10 (4.793) | -5.64 (4.488) | -4.23 (4.723)
Statistical Analysis 1: Comparison: Placebo vs ND-L02-s0201 45 mg; Test type: Superiority; p = 0.668, random coefficient model; Median Difference (Final Values) = -3.16, 95% CI 2-sided [-17.59 to 11.28]
Statistical Analysis 2: Comparison: Placebo vs ND-L02-s0201 90 mg; Test type: Superiority; p = 0.821, random coefficient model; Median Difference (Final Values) = -1.72, 95% CI 2-sided [-16.57 to 13.13]

6. Secondary Outcome: Absolute and Relative Change in ppFVC (%) From Baseline to Week 24
Description: Absolute and Relative Change in ppFVC (%) from Baseline to Week 24. The intent-to-treat population (any randomized participants with treatment assignment according to the planned randomization) is presented.
  ppFVC = percent predicted forced vital capacity
Time Frame: Baseline to Week 24
Population: ITT Population (include any randomized participants with treatment assignment according to the planned randomization)
Measure: Least Squares Mean (Standard Error); unit: percent
Arm/Group | Placebo | ND-L02-s0201 45 mg | ND-L02-s0201 90 mg
Number analyzed (Participants) | 42 | 41 | 40
percent
  Baseline ppFVC | 74.5701 (2.54894) | 79.8896 (2.57837) | 77.2260 (2.60623)
  Week 24 ppFVC | 72.2552 (2.58376) | 75.3849 (2.63382) | 73.9607 (2.65995)
  Change from Baseline to Week 24 in ppFVC | -2.3149 (0.89678) | -4.5046 (0.96141) | -3.2652 (0.96873)
Statistical Analysis 1: Comparison: Placebo vs ND-L02-s0201 45 mg; Change from baseline to Week 24 in ppFVC; Test type: Superiority; p = 0.098, random coefficient model; Median Difference (Final Values) = -2.1897, 95% CI 2-sided [-4.7869 to 0.4075]
Statistical Analysis 2: Comparison: Placebo vs ND-L02-s0201 90 mg; Change from Baseline to Week 24 in ppFVC; Test type: Superiority; p = 0.473, random coefficient model; Median Difference (Final Values) = -0.9503, 95% CI 2-sided [-3.5579 to 1.6573]

7. Secondary Outcome: Percent Change in ppFVC From Baseline to Week 24
Description: Percent Change in ppFVC from Baseline to Week 24. The intent-to-treat population (any randomized participants with treatment assignment according to the planned randomization) is presented.
  ppFVC = percent predicted forced vital capacity
Time Frame: Baseline to Week 24
Population: ITT Population (include any randomized participants with treatment assignment according to the planned randomization)
Measure: Least Squares Mean (Standard Error); unit: percentage
Arm/Group | Placebo | ND-L02-s0201 45 mg | ND-L02-s0201 90 mg
Number analyzed (Participants) | 42 | 41 | 40
percentage | -3.10 (4.793) | -5.64 (4.488) | -4.23 (4.723)
Statistical Analysis 1: Comparison: Placebo vs ND-L02-s0201 45 mg; Test type: Superiority; p = 0.700, random coefficient model; Median Difference (Final Values) = -2.53, 95% CI 2-sided [-15.40 to 10.34]
Statistical Analysis 2: Comparison: Placebo vs ND-L02-s0201 90 mg; Test type: Superiority; p = 0.867, random coefficient model; Median Difference (Final Values) = -1.12, 95% CI 2-sided [-14.31 to 12.07]

8. Secondary Outcome: Summary of Study Treatment Response of FVC
Description: Proportion of participants with an FVC response defined as either having improvement or a decline by 0 to less than or equal to 5%, more than 5% to less than or equal to 10%, and more than 10% at Visit 14 (Day 169).
  Participants with an FVC response were defined as improvement in FVC (ie, FVC value higher than baseline) or a decline of less than or equal to 10% from baseline.
  The intent-to-treat population (any randomized participants with treatment assignment according to the planned randomization) is presented.
  FVC = forced vital capacity
Time Frame: Baseline to Visit 14 (Day 169)
Population: ITT Population (include any randomized participants with treatment assignment according to the planned randomization) with FVC assessment at Visit 14
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | ND-L02-s0201 45 mg | ND-L02-s0201 90 mg
Number analyzed (Participants) | 42 | 41 | 40
Participants
  Improvement | 9 | 7 | 5
  Decline ≥0% to ≤5% | 10 | 6 | 10
  Decline >5% to ≤10% | 8 | 6 | 6
  Decline >10% | 3 | 7 | 4
  Test not done | 12 | 15 | 15

9. Secondary Outcome: Summary of Study Treatment Response of ppFVC
Description: Proportion of participants with an ppFVC response defined as either having improvement or a decline by 0 to less than or equal to 5%, greater than 5% to less than or equal to 10%, and greater than 10% at Visit 14 (Day 169).
  Participants with an ppFVC response were defined as improvement in ppFVC (ie, ppFVC value higher than baseline) or a decline of less than or equal to 10% from baseline.
  The intent-to-treat population (any randomized participants with treatment assignment according to the planned randomization) is presented.
  ppFVC = percent predicted forced vital capacity
Time Frame: Baseline to Visit 14 (Day 169)
Population: ITT Population (include any randomized participants with treatment assignment according to the planned randomization) with ppFVC assessment at Visit 14
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | ND-L02-s0201 45 mg | ND-L02-s0201 90 mg
Number analyzed (Participants) | 42 | 41 | 40
Participants
  Improvement | 9 | 7 | 5
  Decline ≥0% to ≤5% | 10 | 6 | 10
  Decline >5% to ≤10% | 8 | 6 | 6
  Decline >10% | 3 | 7 | 4
  Test not done | 12 | 15 | 15

10. Secondary Outcome: Change in DLCO and DLCO Corrected for Hemoglobin From Baseline to Week 24
Description: Change in diffusion capacity of the lung for carbon monoxide (DLCO) and DLCO corrected for hemoglobin (mL/min/mmHg) from Baseline to Week 24.
  The intent-to-treat population (any randomized participants with treatment assignment according to the planned randomization) is presented.
Time Frame: Baseline to Week 24
Population: ITT Population (include any randomized participants with treatment assignment according to the planned randomization)
Measure: Least Squares Mean (Standard Error); unit: mL/min/mmHg
Arm/Group | Placebo | ND-L02-s0201 45 mg | ND-L02-s0201 90 mg
Number analyzed (Participants) | 42 | 41 | 40
mL/min/mmHg
  Baseline DLCO Corrected for Hemoglobin (mL/min/mmHg) | 12.6709 (0.56489) | 13.0723 (0.57141) | 12.4800 (0.57759)
  Week 24 DLCO Corrected for Hemoglobin (mL/min/mmHg) | 11.7541 (0.58748) | 12.3015 (0.59845) | 12.2669 (0.60460)
  Change from Baseline to Week 24 in DLCO Corrected for Hemoglobin (mL/min/mmHg) | -0.9169 (0.26950) | -0.7708 (0.28085) | -0.2131 (0.28408)
  Baseline DLCO Not Corrected for Hemoglobin (mL/min/mmHg) | 12.4411 (0.55897) | 12.9860 (0.56543) | 12.3792 (0.57155)
  Week 24 DLCO Not Corrected for Hemoglobin (mL/min/mmHg) | 11.5720 (0.57137) | 12.2308 (0.58226) | 12.0661 (0.58804)
  Change from Baseline to Week 24 in DLCO Not Corrected for Hemoglobin (mL/min/mmHg) | -0.8691 (0.26307) | -0.7551 (0.27406) | -0.3131 (0.27721)
Statistical Analysis 1: Comparison: Placebo vs ND-L02-s0201 45 mg; Change from Baseline to Week 24 in DLCO Corrected for Hemoglobin (mL/min/mmHg) in the 45 mg cohort versus placebo; Test type: Superiority; p = 0.708, random coefficient; Mean Difference (Final Values) = 0.1460, 95% CI 2-sided [-0.6226 to 0.9147]
Statistical Analysis 2: Comparison: Placebo vs ND-L02-s0201 90 mg; Change from Baseline to Week 24 in DLCO Corrected for Hemoglobin (mL/min/mmHg) in the 90 mg cohort versus placebo; Test type: Superiority; p = 0.074, random coefficient; Mean Difference (Final Values) = 0.7038, 95% CI 2-sided [-0.0695 to 1.4771]
Statistical Analysis 3: Comparison: Placebo vs ND-L02-s0201 45 mg; Change from Baseline to Week 24 in DLCO Not Corrected for Hemoglobin (mL/min/mmHg) in the 45 mg cohort versus placebo; Test type: Superiority; p = 0.765, random coefficient model; Mean Difference (Final Values) = 0.1140, 95% CI 2-sided [-0.6362 to 0.8641]
Statistical Analysis 4: Comparison: Placebo vs ND-L02-s0201 90 mg; Change from Baseline to Week 24 in DLCO Not Corrected for Hemoglobin (mL/min/mmHg) in the 90 mg cohort versus placebo; Test type: Superiority; p = 0.148, random coefficient model; Mean Difference (Final Values) = 0.5560, 95% CI 2-sided [-0.1986 to 1.3107]

11. Secondary Outcome: Quantitative Changes of Interstitial Lung Abnormalities as Measured by HRCT
Description: Changes of interstitial lung abnormalities as measured by high-resolution computed tomography (HRCT; ie, change in parenchymal feature [Baseline to Week 24]), as determined by qualitative assessment (central radiologist) and quantitative analysis (Quantitative Lung Fibrosis - QLF analysis).
  Quantitative HRCT parameters included the following:
  * Quantitative Lung Fibrosis (QLF) score (% of whole lung field volume)
  * Ground glass opacity (GGO) (% of whole lung field volume)
  * Reticulation (% of whole lung field volume)
  * Honeycombing (% of whole lung field volume)
  * Normal lung (% of whole lung field volume)
  * Emphysema (low attenuation area [LAA]; % of whole lung field volume)
  The intent-to-treat population (any randomized participants with treatment assignment according to the planned randomization) is presented.
Time Frame: Baseline to Week 24
Population: ITT Population (include any randomized participants with treatment assignment according to the planned randomization)
Measure: Least Squares Mean (Standard Error); unit: percentage
Arm/Group | Placebo | ND-L02-s0201 45 mg | ND-L02-s0201 90 mg
Number analyzed (Participants) | 42 | 41 | 40
percentage
  Baseline QLF Score (% of whole lung field volume) | 33.59 (2.189) | 27.45 (2.441) | 27.22 (2.249)
  Week 24 QLF Score (% of whole lung field volume) | 35.87 (2.195) | 29.24 (2.447) | 30.89 (2.258)
  Change from Baseline to Week 24 in QLF Score (% of whole lung field volume) | 2.28 (1.080) | 1.79 (1.194) | 3.67 (1.112)
  Baseline Ground Glass Opacity (% of whole lung field volume) | 5.01 (0.357) | 4.91 (0.399) | 4.72 (0.367)
  Week 24 Ground Glass Opacity (% of whole lung field volume) | 4.77 (0.358) | 4.49 (0.400) | 4.52 (0.369)
  Change from Baseline to Week 24 in Ground Glass Opacity (% of whole lung field volume) | -0.23 (0.177) | -0.41 (0.195) | -0.20 (0.182)
  Baseline Reticulation (% of whole lung field volume) | 27.46 (1.890) | 23.69 (2.108) | 24.03 (1.943)
  Week 24 Reticulation (% of whole lung field volume) | 28.13 (2.001) | 24.97 (2.231) | 26.34 (2.062)
  Change from Baseline to Week 24 in Reticulation (% of whole lung field volume) | 0.67 (0.964) | 1.28 (1.069) | 2.32 (1.010)
  Baseline Honeycombing (% of whole lung field volume) | 4.54 (0.861) | 2.50 (0.961) | 1.54 (0.886)
  Week 24 Honeycombing (% of whole lung field volume) | 6.36 (1.018) | 3.11 (1.135) | 2.37 (1.047)
  Change from Baseline to Week 24 in Honeycombing (% of whole lung field volume) | 1.81 (0.542) | 0.61 (0.604) | 0.83 (0.558)
  Baseline Normal Lung (% of whole lung field volume) | 58.47 (2.281) | 64.52 (2.544) | 65.57 (2.343)
  Week 24 Normal Lung (% of whole lung field volume) | 56.42 (2.287) | 63.35 (2.549) | 62.68 (2.352)
  Change from Baseline to Week 24 in Estimation of Normal Lung (% of whole lung field volume) | -2.05 (1.027) | -1.17 (1.134) | -2.88 (1.057)
  Baseline Emphysema (% of whole lung field volume) | 9.62 (1.640) | 10.66 (1.829) | 8.14 (1.684)
  Week 24 Emphysema (% of whole lung field volume) | 12.08 (1.646) | 9.54 (1.835) | 8.45 (1.694)
  Change from Baseline to Week 24 in Estimation of Emphysema (% of whole lung field volume) | 2.46 (0.936) | -1.12 (1.034) | 0.31 (0.964)
Statistical Analysis 1: Comparison: Placebo vs ND-L02-s0201 45 mg; Change from Baseline to Week 24 in QLF Score (% of whole lung field volume) in the 45 mg cohort versus placebo; Test type: Superiority; p = 0.765, random coefficient model; Mean Difference (Final Values) = -0.48, 95% CI 2-sided [-3.68 to 2.71]
Statistical Analysis 2: Comparison: Placebo vs ND-L02-s0201 90 mg; Change from Baseline to Week 24 in QLF Score (% of whole lung field volume) in the 90 mg cohort versus placebo; Test type: Superiority; p = 0.370, random coefficient model; Mean Difference (Final Values) = 1.40, 95% CI 2-sided [-1.68 to 4.47]
Statistical Analysis 3: Comparison: Placebo vs ND-L02-s0201 45 mg; Change from Baseline to Week 24 in Ground Glass Opacity (% of whole lung field volume) in the 45 mg cohort versus placebo; Test type: Superiority; p = 0.499, random coefficient model; Mean Difference (Final Values) = -0.18, 95% CI 2-sided [-0.70 to 0.34]
Statistical Analysis 4: Comparison: Placebo vs ND-L02-s0201 90 mg; Change from Baseline to Week 24 in Ground Glass Opacity (% of whole lung field volume) in the 90 mg cohort versus placebo; Test type: Superiority; p = 0.901, random coefficient model; Mean Difference (Final Values) = 0.03, 95% CI 2-sided [-0.47 to 0.54]
Statistical Analysis 5: Comparison: Placebo vs ND-L02-s0201 45 mg; Change from Baseline to Week 24 in Reticulation (% of whole lung field volume) in the 45 mg cohort versus placebo; Test type: Superiority; p = 0.676, random coefficient model; Mean Difference (Final Values) = 0.60, 95% CI 2-sided [-2.25 to 3.46]
Statistical Analysis 6: Comparison: Placebo vs ND-L02-s0201 90 mg; Change from Baseline to Week 24 in Reticulation (% of whole lung field volume) in the 90 mg cohort versus placebo; Test type: Superiority; p = 0.242, random coefficient model; Mean Difference (Final Values) = 1.64, 95% CI 2-sided [-1.13 to 4.42]
Statistical Analysis 7: Comparison: Placebo vs ND-L02-s0201 45 mg; Change from Baseline to Week 24 in Honeycombing (% of whole lung field volume) in the 45 mg cohort versus placebo; Test type: Superiority; p = 0.140, random coefficient model; Mean Difference (Final Values) = -1.21, 95% CI 2-sided [-2.82 to 0.40]
Statistical Analysis 8: Comparison: Placebo vs ND-L02-s0201 90 mg; Change from Baseline to Week 24 in Honeycombing (% of whole lung field volume) in the 90 mg cohort versus placebo; Test type: Superiority; p = 0.211, random coefficient model; Mean Difference (Final Values) = -0.98, 95% CI 2-sided [-2.53 to 0.56]
Statistical Analysis 9: Comparison: Placebo vs ND-L02-s0201 45 mg; Change from Baseline to Week 24 in Normal Lung (% of whole lung field volume) in the 45 mg cohort versus placebo; Test type: Superiority; p = 0.568, random coefficient model; Mean Difference (Final Values) = 0.88, 95% CI 2-sided [-2.16 to 3.91]
Statistical Analysis 10: Comparison: Placebo vs ND-L02-s0201 90 mg; Change from Baseline to Week 24 in Normal Lung (% of whole lung field volume) in the 90 mg cohort versus placebo; Test type: Superiority; p = 0.573, random coefficient model; Mean Difference (Final Values) = -0.83, 95% CI 2-sided [-3.76 to 2.09]
Statistical Analysis 11: Comparison: Placebo vs ND-L02-s0201 45 mg; Change from Baseline to Week 24 in Emphysema (% of whole lung field volume) in the 45 mg cohort versus placebo; Test type: Superiority; p = 0.012, random coefficient model; Mean Difference (Final Values) = -3.58, 95% CI 2-sided [-6.35 to -0.81]
Statistical Analysis 12: Comparison: Placebo vs ND-L02-s0201 90 mg; Change from Baseline to Week 24 in Emphysema (% of whole lung field volume) in the 90 mg cohort versus placebo; Test type: Superiority; p = 0.112, random coefficient model; Mean Difference (Final Values) = -2.16, 95% CI 2-sided [-4.82 to 0.51]

12. Secondary Outcome: Qualitative Changes of Interstitial Lung Abnormalities as Measured by HRCT
Description: Changes of interstitial lung abnormalities as measured by high-resolution computed tomography (HRCT; ie, change in parenchymal feature [Baseline to Visit 14 (Day 169)]), as determined by qualitative assessment (central radiologist). The Likert scale values are included in the descriptions presented.
  The intent-to-treat population (any randomized participants with treatment assignment according to the planned randomization) with HRCT assessment at Visit 14/Early Termination is presented.
Time Frame: Baseline to Visit 14 (Day 169)
Population: ITT Population (include any randomized participants with treatment assignment according to the planned randomization) with HRCT assessment at Visit 14/Early Termination
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | ND-L02-s0201 45 mg | ND-L02-s0201 90 mg
Number analyzed (Participants) | 37 | 30 | 34
Participants
  Much better (5) | 0 | 0 | 0
  Better (4) | 0 | 0 | 1
  Same (3) | 28 | 26 | 28
  Worse (2) | 6 | 3 | 3
  Much worse (1) | 3 | 1 | 2
  Unknown | 0 | 0 | 0
Statistical Analysis 1: Comparison: Placebo vs ND-L02-s0201 45 mg; Test type: Superiority; p = 0.256, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo vs ND-L02-s0201 90 mg; Test type: Superiority; p = 0.241, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: Events of IPF Exacerbation or Death and Rate of First IPF Exacerbation
Description: Total number of events of participants who experienced idiopathic pulmonary fibrosis (IPF) exacerbation (ie, an unexplained worsening of dyspnea, evidence of hypoxemia as defined by worsened or severely impaired gas exchange, new radiographic alveolar infiltrates, and an absence of an alternative explanation such as infection, pulmonary embolism, pneumothorax, or heart failure) or death (weeks).
Time Frame: Baseline to study completion, up to Day 239
Population: ITT Population (include any randomized participants with treatment assignment according to the planned randomization)
Measure: Number; unit: events
Arm/Group | Placebo | ND-L02-s0201 45 mg | ND-L02-s0201 90 mg
Number analyzed (Participants) | 42 | 41 | 40
events | 7 | 3 | 4
Statistical Analysis 1: Comparison: Placebo vs ND-L02-s0201 45 mg; Time to First IPF Exacerbation or Death (weeks) in the 45 mg cohort versus placebo; Test type: Superiority; p = 0.517, Log Rank; Hazard Ratio (HR) = 0.649, 95% CI 2-sided [0.189 to 2.225]
Statistical Analysis 2: Comparison: Placebo vs ND-L02-s0201 90 mg; Time to First IPF Exacerbation or Death (weeks) in the 90 mg cohort versus placebo; Test type: Superiority; p = 0.506, Log Rank; Hazard Ratio (HR) = 0.678, 95% CI 2-sided [0.198 to 2.324]
Statistical Analysis 3: Comparison: Placebo vs ND-L02-s0201 45 mg; Rate of First IPF Exacerbation (%) in the 45 mg cohort versus placebo; Test type: Superiority; p = 0.313, Fisher Exact; Proportion Difference (Final Values) = -9.3, 95% CI 2-sided [-25.2 to 5.5] — The 95% Confidence Interval for difference in proportions are based on the Chan-Zhang method
Statistical Analysis 4: Comparison: Placebo vs ND-L02-s0201 90 mg; Rate of First IPF Exacerbation (%) in the 90 mg cohort versus placebo; Test type: Superiority — The 95% Confidence Interval for difference in proportions are based on the Chan-Zhang method; p = 0.376, Chi-squared; Proportion Difference (Final Values) = -6.7, 95% CI 2-sided [-22.6 to 9.2]

14. Secondary Outcome: Events of Hospitalization for Respiratory Ailments or Death
Description: Events (participants who experienced hospitalization for respiratory ailments or died) for respiratory ailments are presented.
  The intent-to-treat population (any randomized participants with treatment assignment according to the planned randomization) is presented.
Time Frame: up to 12 weeks after the end of study treatment
Population: ITT Population (include any randomized participants with treatment assignment according to the planned randomization)
Measure: Number; unit: events
Arm/Group | Placebo | ND-L02-s0201 45 mg | ND-L02-s0201 90 mg
Number analyzed (Participants) | 42 | 41 | 40
events | 5 | 3 | 3
Statistical Analysis 1: Comparison: Placebo vs ND-L02-s0201 45 mg; Rate of Hospitalization for Respiratory Ailments (%) in the 45 mg cohort versus placebo; Test type: Superiority; p = 0.713, Fisher Exact; Proportion Difference (Final Values) = -4.6, 95% CI 2-sided [-19.2 to 9.6] — The 95% Confidence Interval for difference in proportions are based on the Chan-Zhang method
Statistical Analysis 2: Comparison: Placebo vs ND-L02-s0201 90 mg; Rate of Hospitalization for Respiratory Ailments (%) in the 90 mg cohort versus placebo; Test type: Superiority; p = 0.713, Fisher Exact; Proportion Difference (Final Values) = -4.4, 95% CI 2-sided [-19.2 to 10.7] — The 95% Confidence Interval for difference in proportions are based on the Chan-Zhang method

15. Secondary Outcome: Total Events of Death Due to All Causes
Description: Rate of mortality due to all causes is presented. Overall survival was defined as the time from start of study treatment to death due to any cause.
Time Frame: up to 12 weeks after the end of study treatment
Population: ITT Population (include any randomized participants with treatment assignment according to the planned randomization)
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | ND-L02-s0201 45 mg | ND-L02-s0201 90 mg
Number analyzed (Participants) | 42 | 41 | 40
Participants | 1 | 1 | 0
Statistical Analysis 1: Comparison: Placebo vs ND-L02-s0201 45 mg; Overall Survival (weeks) in the 45 mg cohort versus placebo; Test type: Superiority; p = 0.937, Log Rank
Statistical Analysis 2: Comparison: Placebo vs ND-L02-s0201 90 mg; Overall Survival (weeks) in the 90 mg cohort versus placebo; Test type: Superiority; p = 0.414, Log Rank
Statistical Analysis 3: Comparison: Placebo vs ND-L02-s0201 45 mg; Rate of Mortality (%) in the 45 mg cohort versus placebo; Test type: Superiority; p > 0.999, Fisher Exact; Proportion Difference (Final Values) = 0.1, 95% CI 2-sided [-10.4 to 10.9] — The 95% Confidence Interval for difference in proportions are based on the Chan-Zhang method
Statistical Analysis 4: Comparison: Placebo vs ND-L02-s0201 90 mg; Rate of Mortality (%) in the 90 mg cohort versus placebo; Test type: Superiority; p > 0.999, Fisher Exact; Proportion Difference (Final Values) = -2.4, 95% CI 2-sided [-13.1 to 6.8] — The 95% Confidence Interval for difference in proportions are based on the Chan-Zhang method

16. Secondary Outcome: Events of Deterioration of IPF Resulting in Lung Transplantation or Death and Rate of Deterioration of IPF Resulting in Lung Transplantation
Description: Events of deterioration of Idiopathic Pulmonary Fibrosis (IPF) resulting in lung transplantation (LP; up to 12 weeks after the end of study treatment) or death (weeks) and rate of deterioration of IPF resulting in lung transplantation (up to 12 weeks after the end of study treatment) are presented.
  Total events = Participants who experience deterioration of IPF resulting in LP (or died).
  Rate of Deterioration = Rate of Deterioration of IPF Resulting in LP.
Time Frame: Baseline to 12 weeks after end of study treatment
Population: ITT Population (include any randomized participants with treatment assignment according to the planned randomization)
Measure: Number; unit: events
Arm/Group | Placebo | ND-L02-s0201 45 mg | ND-L02-s0201 90 mg
Number analyzed (Participants) | 42 | 41 | 40
events
  Total events to Deterioration of IPF Resulting in LP or Death: | 3 | 1 | 0
  Rate of Deterioration of IPF Resulting in LP: Total Events | 2 | 0 | 0
Statistical Analysis 1: Comparison: Placebo vs ND-L02-s0201 45 mg; Rate of Deterioration of IPF Resulting in Lung Transplantation (%) in the 45 mg cohort versus placebo; Test type: Superiority; p = 0.494, Fisher Exact; Proportion Difference (Final Values) = -4.8, 95% CI 2-sided [-16.6 to 4.6] — The 95% Confidence Interval for difference in proportions are based on the Chan-Zhang method
Statistical Analysis 2: Comparison: Placebo vs ND-L02-s0201 90 mg; Rate of Deterioration of IPF Resulting in Lung Transplantation (%) in the 90 mg cohort versus placebo; Test type: Superiority; p = 0.494, Fisher Exact; Proportion Difference (Final Values) = -4.8, 95% CI 2-sided [-16.2 to 4.5] — The 95% Confidence Interval for difference in proportions are based on the Chan-Zhang method

ADVERSE EVENTS:
Time Frame: Approximately 40 weeks (from screening to follow-up visit).
Description: Safety population includes all participants who received at least one dose of study treatment.
Groups:
- Placebo: Intravenous placebo infusion every 2 weeks (plus/minus 4 days for Visit 3 or plus/minus 7 days for Visits 4 to 13, ensuring a minimum of 7 days between each dose) for a total of 12 doses.
- ND-L02-s0201 45 mg: ND-L02-s0201: 45 mg intravenous administration every 2 weeks (plus/minus 4 days for Visit 3 or plus/minus 7 days for Visits 4 to 13, ensuring a minimum of 7 days between each dose) for a total of 12 doses
- ND-L02-s0201 90 mg: ND-L02-s0201: 90 mg intravenous administration every 2 weeks (plus/minus 4 days for Visit 3 or plus/minus 7 days for Visits 4 to 13, ensuring a minimum of 7 days between each dose) for a total of 12 doses.
Arm/Group | Placebo | ND-L02-s0201 45 mg | ND-L02-s0201 90 mg
All-Cause Mortality (participants affected / at risk) | 1/42 | 1/41 | 0/40
Serious Adverse Events (participants affected / at risk) | 9/42 | 4/41 | 6/40
Other Adverse Events (participants affected / at risk) | 35/42 | 37/41 | 37/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=42) | ND-L02-s0201 45 mg (N=41) | ND-L02-s0201 90 mg (N=40)
Cervical radiculopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Anastomotic haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Thalamic infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Vascular stent stenosis (General disorders) | 0 (0) | 0 (0) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=42) | ND-L02-s0201 45 mg (N=41) | ND-L02-s0201 90 mg (N=40)
Vision blurred (Eye disorders) | 0 (0) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (5) | 2 (2) | 1 (2)
Nausea (Gastrointestinal disorders) | 2 (2) | 4 (4) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 3 (3)
Fatigue (General disorders) | 3 (3) | 3 (3) | 5 (5)
Infusion site reaction (General disorders) | 1 (1) | 6 (6) | 2 (3)
Oedema peripheral (General disorders) | 1 (1) | 1 (1) | 2 (2)
Pain (General disorders) | 2 (2) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0) | 2 (2)
Sinusitis (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 9 (12) | 4 (4) | 6 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (7) | 4 (4) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 0 (0) | 0 (0)
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 3 (3) | 4 (4)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 3 (3)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1) | 3 (3)
Lipase increased (Investigations) | 0 (0) | 2 (2) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 3 (4) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 3 (4) | 14 (46) | 19 (56)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 4 (7) | 3 (3)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 3 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3) | 3 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2)
COVID-19 (Infections and infestations) | 2 (2) | 1 (1) | 3 (3)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 0 (0) | 3 (3) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 2 (2) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (3) | 1 (2) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Nitto Denko Corporation agreements with investigators vary; constant is Nitto's right to embargo communications regarding trial results prior to public release for a period <30 days from submittal for review. Nitto will not prohibit investigators from publishing but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2020-06-17): https://cdn.clinicaltrials.gov/large-docs/01/NCT03538301/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-13): https://cdn.clinicaltrials.gov/large-docs/01/NCT03538301/SAP_001.pdf